CLINICAL TRIAL: NCT06641869
Title: A 12-week , Randomized, Open-label Study of PCC1 in Healthy Volunteers for Skin Rejuvenation
Brief Title: Study of PCC1 for Skin Rejuvenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Express Rx, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EXRX023
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Skin Rejuvenation
MeSH Terms: interventions — procyanidin trimer C1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- PCC1 Group (Experimental): Dosage Form: Oral dietary supplement. Dosage: 2.5 mg of procyanidin C1. Frequency: Administered once daily. Duration: 12 weeks.
  Interventions: Dietary Supplement: procyanidin C1
- Placebo (Placebo Comparator): Dosage Form: Oral placebo supplement. Dosage: Administered once daily. Duration: 12 weeks.
  Interventions: Dietary Supplement: Placebo
- PCC1 Complex (Experimental): Dosage: 5 mg of procyanidin C1. Frequency: Administered once daily. Duration: 12 weeks.
  Interventions: Dietary Supplement: PCC1 complex

INTERVENTIONS:
Dietary Supplement: procyanidin C1 — Proprietarily extracted procyanidin C1
  Arms: PCC1 Group
Dietary Supplement: Placebo — Placebo
  Arms: Placebo
Dietary Supplement: PCC1 complex — 5 mg of procyanidin C1. Frequency: Administered once daily. Duration: 12 weeks.
  Arms: PCC1 Complex

SUMMARY:
This clinical trial will assess the efficacy of PCC1 for skin rejuvenation. The primary objective is to determine whether these interventions enhance skin barrier function, reduce wrinkles, and improve skin texture and radiance over a 12-week period. The study will involve healthy participants applying the treatments and undergoing assessments at baseline, 6 weeks, and 12 weeks. Secondary objectives include evaluating the safety and tolerability of PCC1, with any adverse effects closely monitored during the trial.

DETAILED DESCRIPTION:
As skin ages, intrinsic and extrinsic factors contribute to cellular senescence, disrupting the skin's structure and function. Senescent cells accumulate in the skin, leading to the secretion of senescence-associated secretory phenotype (SASP) factors, which promote inflammation and degrade extracellular matrix proteins like collagen. These changes result in wrinkles, loss of elasticity, and reduced skin barrier function. The study explores anti-senescence strategies using senolytic agents that selectively eliminate senescent cells, aiming to rejuvenate the skin. Compounds like PCC1 and Cellumiva have shown promise in targeting senescent cells by inducing apoptosis and reducing SASP expression, offering a novel approach to skin aging therapy.

This clinical trial is designed to evaluate the efficacy and safety of PCC1 in skin rejuvenation over 12 weeks. Healthy female participants aged 45-65 will be randomly assigned to receive PCC1 or a placebo. The study will measure skin barrier function, wrinkle reduction, and texture/radiance improvements using imaging technologies and participant feedback. Safety will also be monitored through adverse event reporting.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 45-65
* any skin type according to the Glogau scale
* No significant underlying health conditions affecting skin.
* Willingness to comply with the study protocol.
* Capacity to personally give informed consent (consent via legally authorized representative will not be accepted) and who are willing to comply with all study-related procedures and assessments;

Exclusion Criteria:

* Presence of any dermatological conditions or use of retinoids or similar compounds within 6 months of the study.
* patients with active skin diseases (e.g. atopic dermatitis, psoriasis, rosacea, seborrheic dermatitis)
* patients using other anti-aging treatments within 1 month

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 74 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-08-10 (Actual)

PRIMARY OUTCOMES:
Skin Barrier Function | at baseline, week 6, and week 12.
  Measured via Trans-Epidermal Water Loss (TEWL) using a VapoMeter at baseline, week 6, and week 12.
Wrinkle Reduction | at baseline, week 6, and week 12.
  Quantified using Antera 3D imaging analysis for wrinkle indentation.
Skin Texture and Radiance | at baseline, week 6, and week 12.
  Evaluated via VISIA-CR imaging and expert clinical grading

SECONDARY OUTCOMES:
Self-Perceived Skin Improvements | 12 weeks
  This outcome will be assessed using the Self-Perceived Skin Improvement Scale (SPSIS), a questionnaire with a minimum score of 0 and a maximum of 100. Higher scores indicate better self-perceived skin improvements. Participants will evaluate hydration, smoothness, radiance, and overall appearance of their skin. Results will be measured at baseline and at the end of 12 weeks. Separate outcome measures will be reported for each parameter (hydration, smoothness, radiance), based on individual scores from the SPSIS.
Safety and Tolerability | 12 weeks
  Monitored through adverse event reports, particularly any irritation or dermatological reactions

CONTACTS AND LOCATIONS:
Overall Officials: Emilia Loewe, Principal Investigator — Express Rx, Inc
Locations (1):
- University of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided